CLINICAL TRIAL: NCT04253184
Title: Micra AV Transcatheter Pacing System Post-Approval Registry
Acronym: Micra AV PAS
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Micra AV PAS
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Micra AV Transcatheter Pacing System — The Micra AV Transcatheter Pacing System (TPS) is a miniaturized single chamber pacemaker that is delivered via catheter through the femoral vein and is implanted directly inside the right ventricle of the heart to provide bipolar sensing and pacing. The Micra AV system provides a form of VDD pacing that is based on mechanical atrial sensing utilizing a 3-axis accelerometer.

SUMMARY:
Medtronic is sponsoring the Micra AV Registry using the Micra AV system for continued surveillance of chronic atrioventricular synchronous pacing as intended, through the collection of data based on routine clinical care practice, following commercial release.

The Micra AV Registry is conducted within Medtronic's Product Surveillance Registry (PSR) platform.

DETAILED DESCRIPTION:
The Micra AV Registry is a global, prospective, observational, multi-site registry. Patients enrolled in the Micra AV Registry will be prospectively followed for a minimum of 3 years post-implant or until registry closure, patient death, patient exit from the registry (i.e., withdrawal of consent).

Enrolled patients will have scheduled follow-up visits at least annually or as prompted by reportable adverse events; however, all Micra AV system follow-up patient visits are to be reported. Therefore, if more frequent scheduled visits occur per a provider's routine clinical care practice, those visits are reported. The total estimated registry duration is 4.5 years

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient is intended to receive or be treated with a Micra AV Transcatheter Pacing System and must be enrolled prior to the implant procedure

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients intended to be implanted with a Micra AV system are eligible for enrollment and all patients must be consented prior to the implant. As such, only geographies with regulatory approval for the Micra system are eligible to enroll patients (see locations section).
  All patients enrolled and successfully implanted with a Micra AV system will be followed for a minimum of 3 years, unless a patient is exited from the registry due to an unavoidable reason. If a Micra AV system is not successfully implanted, patients will be exited from the registry unless a Micra AV System and/or implant procedure related event is identified, for which the patient will be followed until the event is resolved or no further actions need to be taken.
Sampling Method: Non-Probability Sample
Enrollment: 802 (Actual)
Dates: Start 2020-02-08 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Rate of pacemaker syndrome | After 3 years of Follow Up
  To characterize the rate of pacemaker syndrome resulting in a system revision at 3-years post-implant.

SECONDARY OUTCOMES:
Acute complication rate | After 30 days of Follow Up
  To estimate the acute major complication rate related to the Micra AV system and/or procedure.
Long-term complication rate | After 3 years of Follow up
  To estimate the 3-year major complication rate related to the Micra AV system and/or procedure.

OTHER OUTCOMES:
AV Synchrony Loss | After 3 years of Follow up
  To characterize the rate and severity of adverse events potentially related to AV synchrony loss
System and Procedure Related Adverse Events | After 3 years of Follow up
  Summarize Micra AV system or procedure related adverse events
Implant Characteristics | Up to 3 years of Follow Up
  Characterize the implant procedure
Electrical Performance | After 3 years of Follow up
  Characterize electrical performance over time
A4 Amplitude | After 3 years of Follow up
  Characterize A4 amplitude over time

CONTACTS AND LOCATIONS:
Locations (89):
- United States (46):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Eisenhower Desert Cardiology Center, Rancho Mirage, California
  - Sequoia Hospital, Redwood City, California
  - Yale New Haven Health System, New Haven, Connecticut
  - Baptist Health, Jacksonville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Indiana University Health Methodist Research Institute, Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Saint Elizabeth Healthcare, Edgewood, Kentucky
  - The John Hopkins Hospital, Baltimore, Maryland
  - MedStar Baltimore, Baltimore, Maryland
  - TidalHealth Peninsula Regional Medical Center, Salisbury, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Heart, Ypsilanti, Michigan
  - Metropolitan Cardiology Consultants, Coon Rapids, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Forrest General Hospital, Hattiesburg, Mississippi
  - Saint Lukes Health System, Kansas City, Missouri
  - Monmouth Cardiology, Ocean City, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Northwell Health, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - New York-Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Medicor Associates, Erie, Pennsylvania
  - Lankenau Institute for Medical Research, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Shadyside, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Consultants in Cardiology, Fort Worth, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Brussels
  - UZ Leuven-Campus - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Régional de la Citadelle, Liège
- Canada (4):
  - University of Calgary, Calgary
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal
  - Montreal Heart Institute, Montreal
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
- Na Homolce Hospital, Prague, Czechia
- Odense Universitetshospital, Odense, Denmark
- France (6):
  - CHRU de Tours - Hopital trousseau, Chambray-lès-Tours
  - Centre Hospitalier Universitaire de Clermont-Ferrand-Gabriel-Montpied, Clermont-Ferrand
  - Hôpital Européen Georges-Pompidou, Paris
  - Hôpital Haut-Lévêque - CHU de Bordeaux, Pessac
  - CHU Toulouse - Hôpital Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
- Germany (5):
  - St. Vinzenz-Hospital Köln, Cologne
  - Universitätsklinikum Jena - Friedrich Schiller Universität, Jena
  - Städtisches Klinikum Karlsruhe GmbH, Karlsruhe
  - Robert Bosch Krankenhaus, Stuttgart
  - Klinikum Villingen-Schwenningen, Villingen-Schwenningen
- Hygeia Hospital, Athens, Greece
- Barzilai Medical Center Ashkelon, Ashkelon, Israel
- Italy (4):
  - Azienda Ospedaliera Sepdali Civili di Brescia, Brescia
  - Maria Cecilia Hospital, Cotignola
  - Centro Cardiologico Monzino, Milan
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
- Malaysia (2):
  - Cardiac Vascular Sentral Kuala Lumpur, Kuala Lumpur
  - Institut Jantung Negara, Kuala Lumpur
- Netherlands (2):
  - Amsterdam UMC - Locatie AMC, Amsterdam
  - HagaZiekenhuis - Locatie Leyweg, The Hague
- Akerhus University Hospital, Oslo, Norway
- Centro Hospitalar de Lisboa Ocidental, E.P.E. Hospital de Santa Cruz, Carnaxide, Portugal
- King Salman Heart Center - King Fahad Medical City, Riyadh, Saudi Arabia
- Klinicki Centar Srbije, Belgrade, Serbia
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Spain (3):
  - Hospital Universitario da Coruña, A Coruña
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela
- Switzerland (2):
  - Inselspital-Universitatsspital Bern, Bern
  - UniversitätsSpital Zürich, Zurich
- United Kingdom (3):
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Northampton General Hospital NHS Trust, Northampton
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No